CLINICAL TRIAL: NCT03321123
Title: Adoptive Therapy With MB-CART19.1 in Patients With Relapsed/Refractory CD19-positive B Cell Acute Lymphoblastic Leukemia
Brief Title: MB-CART19.1 in Patients With R/R ALL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Children's Medical Center (Other)
Collaborators: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCMC CART 20170920
Record Dates: First submitted 2017-09-20; First posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Precursor B-Lymphoblastic Lymphoma/Leukaemia Refractory
Keywords: B cell Acute Lymphoblastic Leukemia; relapsed or refractory; CD-19 Positive
MeSH Terms: conditions — Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CRA treatment (Experimental): The drug for this trial is autologous T cells transduced with the lentiviral vector pLTG1563 (MB-CART19.1). The dose is 2x10e6 ~2x10e7 MB-CART19.1/kg.
  A leukapheresis for the patient will be performed for MB-CART19.1 generation. All patients will receive lymphodepleting chemotherapy with fludarabine 30 mg/m2/d intravenously (iv) on days -5,-4,-3 and -2 cyclophosphamide 500 mg/m2/d iv on day -3,-2 before CAR T cell transfer to enhance the in vivo expansion of CAR T cells.
  Interventions: Drug: MB-CART19.1

INTERVENTIONS:
Drug: MB-CART19.1 — Miltenyi Biotec has established a semi-automated manufacturing process that can be made available to academic settings for systematic exploration of CAR strategies in advanced clinical studies. Closed-system operation, improved robustness, simplified work flows, and reduced labor intensity, while maintaining strict adherence to regulatory guidelines, allows for decentralized manufacturing. In this study, we will explore autologous 2nd generation CD19 CAR T cell products in patients with relapsed and refractory disease incurable with standard therapies.
  Other Names: Miltenyi CD-19 CAT-T cell

SUMMARY:
Precursor-B acute lymphoblastic leukemia (ALL) is the most common cancer in childhood. Despite major advances in ALL therapy, 20% of children and 40-50% of adults fail state-of-the art first-line treatment. But there is a strong need for alternative treatments to cure chemotherapy-refractory and relapsed B cell malignancies in pediatric patients. Relapsed and refractory B cell malignancies remain a therapeutic challenge, as these diseases are characterized by adverse survival. These cancers share a cell origin from the B-cell lineage and consequent surface expression of B-lineage markers such as CD19 and CD22. Chimeric antigen receptor (CAR) engineered T cell therapy has recently emerged as a new modality to target B cell malignancies. CARs couple a single-chain Fv (scFv) domain directed against a B-lineage-specific antigen to T-cell activating intracellular signaling domains. CAR gene-modified T cell interaction with target cells occurs in a HLA-independent fashion, so that a single vector can be used to treat all patients with cancers that express the target antigen. Miltenyi Biotec has established a semi-automated manufacturing process that can be made available to academic settings for systematic exploration of CAR strategies in advanced clinical studies. Closed-system operation, improved robustness, simplified work flows, and reduced labor intensity, while maintaining strict adherence to regulatory guidelines, allows for decentralized manufacturing. In the proposed phase II study, the investigator will explore autologous 2nd generation CD19 CAR T cell products in patients with relapsed and refractory disease incurable with standard therapies.

DETAILED DESCRIPTION:
This is an open-label, non-randomized phase II paediatric study. In this study, eligible patients will receive autologous T cells transduced with the lentiviral vector pLTG1563 (MB-CART19.1) at a doesage of 2x10e6 ~2x10e7 CAR-transduced T cells/kg.

Upon enrollment, leukapheresis will be performed for MB-CART19.1 generation. Patients with high disease burden at screening (e.g. ALL with M3 marrow and 10.000/L blasts in peripheral blood) may receive bridging chemotherapy after leukapheresis, to avoid critical tumor lysis syndrome and cytokine release syndrome (CRS) by subsequent lymphodepleting chemotherapy and CAR transfer.

All patients will receive lymphodepleting chemotherapy with fludarabine 30 mg/m2/d intravenously (iv) on days -5,-4,-3 and -2 cyclophosphamide 500 mg/m2/d iv on day -3,-2 before CAR T cell transfer to enhance the in vivo expansion of CAR T cells.

Patients will receive freshly prepared MB-CART19.1 on day 0, corresponding to day 12 (48 hours) of manufacturing, at a dose of 2x10e6 ~2x10e7/kg MB-CART19.1 T cells as defined in the study design section. The appropriate volume for the target cell dose will be drawn up and given as an IV injection over 30 minutes through a large vein peripherally or centrally.

The primary objectives are:

* To assess the safety and tolerability of MB-CART19.1.
* To evaluate the biological activity of adoptive transfer of autologous MB-CART19.1 in patients with R/R CD19-positive B cell lymphoblastic leukemia.

The primary endpoint is Overall response rate (ORR):ORR in ALL patients is defined as the rate of complete remission (CR, CRh) on day 28.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤18 years (if deemed fit by treating investigator)
* CD19 expression must be detected on the malignant cells by flow cytometry.
* Patients with relapsed disease with >5% blasts in BM (M2 or M3) after at least one standard chemotherapy and one salvage regimen who are ineligible for allogeneic stem cell transplant (alloSCT)
* Patients have refractory disease activity precluding alloSCT at this time, or patients who have relapsed post alloSCT at least 100 days post-transplant, with no evidence of active GVHD, and no longer taking immunosuppressive agents for at least 30 days prior to enrollment.
* Patients with combined extramedullary ALL are eligible if extramedullary disease has been successfully cleared by conventional therapy at the time of inclusion (e.g. intrathecal chemotherapy, orchiectomy). This includes patients with combined CNS-2 (<5 WBC/µl CSF, with blasts on cytospin) or CNS-3 (5WBC/µl CSF, with blasts on cytospin) disease and patients with combined testicular relapse.
* Patients and/or parents must give their written informed consent/assent.

Exclusion Criteria:

* Rapidly progressive disease that in the estimation of live less than 12 weeks
* Isolated extramedullary relapse (CNS and/or testicular) in ALL
* Current autoimmune disease, or history of autoimmune disease with potential CNS involvement
* Active clinically significant CNS dysfunction (including but not limited to uncontrolled seizure disorders, cerebrovascular ischemia or hemorrhage, dementia, paralysis)
* History of an additional malignancy other than non-melanoma skin cancer or carcinoma in situ unless disease free for ≥3 years.
* Pulmonary function: Patients with pre-existing severe lung disease (FEV1 or FVC < 65%) or an oxygen requirement of >28% O2 supplementation or active pulmonary infiltrates on chest X-ray at the time scheduled for T cell infusion
* Cardiac function: Fractional shortening <28% or left ventricular ejection fraction <50% by echocardiography
* Renal function: Creatinine clearance <50 mL/min/1.73 m2

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 1 Month
  ORR in ALL patients is defined as the rate of complete remission (CR, CRh) on day 28

SECONDARY OUTCOMES:
Overall incidence and severity of adverse events. | 1 Months
  Overall incidence and severity of adverse events will measure in this trial. Including: 1,Risks related to targeting of CD19+ normal B-cells; 2,Allergic reactions to CAR T cell infusion; 3, Cytokine release syndrome (CRS); 4, neurological toxicities; 5,Risks related to transfer of donor T cells after previous alloSCT; 6, Risks related to lentiviral gene transfer into human cells.
Rate of ALL patients achieving MRD negative CR | 12 Months
  The rate of ALL patients achieving MRD negative CR in D28; 3,6,12months.
Relapse rate and time to relapse | 12 Months
  Overall rate of relapse and the time to relapse from CART cell transfused.

OTHER OUTCOMES:
Disease-free and overall survival at 1 year after adoptive immunotherapy with MB-CART19.1 in patients not receiving alloSCT | 12 Months
  CART treatment is an adoptive immunotherapy, and the CART cells will disaper after infusion. Then the patient relapsed. Allo-SCT can rebuild a new immune system to detec and destory cancer cell.
Level of circulating CAR T cells | 12 Months
  CART treatment is an adoptive immunotherapy, and the CART cells will disaper after infusion. The investigator need to detec the circulating CAR-T cell after infusion regularly.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Chen, MD,PhD, Principal Investigator — Shanghai Children Medicine Center

IPD SHARING:
Plan to Share IPD: Undecided